CLINICAL TRIAL: NCT02474238
Title: Randomized Clinical Trial Comparing Neodynium:Ytrium-aluminium-garnet (Nd:YAG) Laser and Sequential Double Frequency YAG-Nd:YAG Laser Iridotomy in Patients With Dark Iris
Brief Title: Comparing Nd:YAG Laser and Sequential Double Frequency YAG-Nd:YAG Laser Iridotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Weerawat Kiddee, Asst.Prof.Weerawat Kiddee, Prince of Songkla University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EC-58-093-02-1
Record Dates: First submitted 2015-06-11; First posted 2015-06-17 (Estimated); Last update posted 2018-08-27 (Actual); Status verified 2018-08

CONDITIONS: Angle Closure Glaucoma
Keywords: Iridotomy
MeSH Terms: conditions — Glaucoma, Angle-Closure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- The sequential technique (Experimental): By using the double frequency YAG laser to make the initial bore and the Nd:YAG laser to complete the perforation on iris.
  Interventions: Device: The sequential technique
- The pure Nd:YAG laser technique (Active Comparator): By using the pure Nd:YAG to make a complete perforation on iris.
  Interventions: Device: The pure Nd:YAG laser technique

INTERVENTIONS:
Device: The sequential technique — By using 'the double frequency YAG laser' to make the initial bore and 'the Nd:YAG laser' to complete the perforation on iris.
  Arms: The sequential technique
Device: The pure Nd:YAG laser technique — By using 'the pure Nd:YAG laser' to make a complete perforation on iris.
  Arms: The pure Nd:YAG laser technique

SUMMARY:
No single type of laser or set of laser parameters is appropriate for all type of irides. Pure Nd:YAG laser iridotomy is very effective in the light color irides. It was considered as the gold standard for iridotomy. It, however, is less effective and causes some complication such as iris hemorrhage especially in patients with dark iris.

DETAILED DESCRIPTION:
By using the double frequency YAG to make the initial bore and the Nd:YAG laser to complete the perforation, the technique should be able to effectively combine most of the advantages of both lasers whilst avoiding their disadvantages. It is possibly the ideal iridotomy technique to use in the Asian irides. The investigators aim to study the energy use for laser iridotomy comparing between the two techniques as well as objectively measure the variables associated with complications.

ELIGIBILITY:
Inclusion Criteria:

* Patient in need to have a laser iridotomy

  * primary angle closure glaucoma or
  * primary angle closure or
  * primary angle closure suspect (needed repeated pupil dilation) or
  * fellow eyes of acute angle closure crisis, and
* Age of at least 18 years, and
* Dark iris patients (only black and dark brown color)

Exclusion Criteria:

* Eye with acute angle closure crisis
* Active conjunctiva or corneal infection or inflammation
* Active anterior uveitis
* History of any prior laser treatment
* History intraocular surgery
* Eye with corneal scar
* Corneal haziness obscure iridotomy site
* Endothelial cell count less than 1000 cells/mm2 (pre-laser)
* Iris color other than black or dark brown
* Inability to sit at the slit lamp to have laser done

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2015-05; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Laser energy | 1-hour
  Total energy used to create patency on the iris

SECONDARY OUTCOMES:
Bleeding | 1-hour
  iris bleeding immediate after laser reported as Yes or No
Corneal endothelial cell count | 12-month
  Corneal endothelial cell count directly over the area of laser
Central corneal thickness | 12-month
  Central corneal thickness
Patency of iridotomy | 12-month
  Iridotomy patency is confirmed objectively reported as yes or no
Intraocular pressure spike | 1-hour
  Intraocular pressure spike if present mean that IOP evelation of at least 8mmHg from baseline intraocular pressure

CONTACTS AND LOCATIONS:
Overall Officials: Asst.Prof.Weerawat Kiddee, MD, Principal Investigator — Prince of Songkla University
Locations (1):
- Weerawat Kiddee, Hat Yai, Changwat Songkhla, Thailand